CLINICAL TRIAL: NCT04929652
Title: Surufatinib Combine With Immunotherapy and Chemotherapy for Second-line Treatment in Advanced Colorectal Cancer：An-open ，Single-arm，Multic-centers Ⅰb/Ⅱ Study.
Brief Title: Surufatinib Combine With Immunotherapy and Chemotherapy for Second-line Treatment in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Liangjun Zhu M.M., Ward Director of Internal Medicine, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-C102/JS-GI2101
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced CRC (Experimental): Patients with Advanced CRC were given Surufatinib Combine With Immunotherapy and Chemotherapy.
  Interventions: Drug: Surufatinib,Camrelizumab,Irinotecan,GM-CSF

INTERVENTIONS:
Drug: Surufatinib,Camrelizumab,Irinotecan,GM-CSF — 1. Dose climbing stage design (n=12) :
     Surufatinib: Oral, 3w.The initial dose of 250mg/ day (n=6) : If 2 out of 6 patients developed > DLT in the first treatment cycle, the exploratory dose was 200 mg/ day; if ≤2 out of 6 patients developed DLT, the exploratory dose was 300mg/ day (n=6);At the next dose phase, if 2 out of 6 patients with > developed DLT, the previous dose was recommended or the study was terminated;If no more than 2 out of 6 patients developed DLT, the dose was the recommended dose；PD-1,200mg, iv,D1, 3w；Irinotecan: 200mg/㎡, iv, D1, 3w；GM-CSF,D2, D3, D4, D5, D6 and D7 in the first week of each cycle ；
  2. Dose expansion phase design(n=36):
     1. Surufatinib: Oral, 3w. the dose was set according to the recommended dose in the dose climbing stage;
     2. PD-1(Camrelizumab) : 200mg, iv,D1, 3w;
     3. Irinotecan: 200mg/㎡, iv, D1, 3w;
     4. GM-CSF: continuous administration of D2, D3, D4, D5, D6 and D7 in the first week of each cycle, 5ug/kg once per body weight, once a day, 3w.
  Other Names: Chemotherapy(Irinotecan),Immunotherapy(Camrelizumab,GM-CSF)

SUMMARY:
The objective is to investigate the efficacy and safety of Surufatinib Combine With Immunotherapy and Chemotherapy for Second-line Treatment in Advanced Colorectal Cancer.

DETAILED DESCRIPTION:
Currently second-line treatment is the Anti-vascular combined chemotherapy, the third line standard is multi-target antivascular therapy, RIGONIVO research in three line treatment of good data, but failed to further validation in the real world, one of the reasons may be the third line therapy, patients physical score is relatively poor, immunotherapy to join may play a role,As we know, the PS score of all effective cases in the Rigonivo study was 0. Therefore, if the idea of antivascular combined immunotherapy is moved forward, it is possible to achieve better efficacy,Based on the above,The objective is to investigate the efficacy and safety of Surufatinib Combine With Immunotherapy and Chemotherapy for Second-line Treatment in Advanced Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures.
2. Male or female, age18-75 years.
3. Pathologically confirmed unresectable locally advanced or advanced metastatic colorectal cancer .
4. First-line use of oxaliplatin in combination with fluorouracil, whether or not combined with macromolecular targeted agents (Cetuximab or Bevacizumab);
5. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
6. The patient had previously failed standard first-line systemic chemotherapy,Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy(Previous standard treatment did not include small molecule inhibitors of anti-angiogenesis and Immunotherapy for PD-1 and PD-L1).
7. A WHO performance status equal to 0-1 and a minimum life expectancy of 12 weeks.
8. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelet count ≥100×109 / L
   3. Hemoglobin≥9 g/dL
   4. Albumin≥3g/dL
   5. Aspartate aminotransferase (AST) ≤ 2.5 × ULN if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
   6. Total bilirubin (TBL)≤ 1.5 × ULN if no liver metastases or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   7. Creatinine≤ 1.5 × ULN concurrent with creatinine clearance ≤50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is ≤1.5 × ULN.
9. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

   1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation. Male patients should be willing to use barrier contraception (i.e., condoms).
   3. For inclusion in study, patient must provide a written informed consent.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior treatment with Surufatinib and other small molecule antiangiogenic targeted drug therapy;.
   2. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   3. Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
   4. First line treatment with irinotecan.
   5. Previous experience with other anti-PD-1 antibody therapy or other PD-L1 immunotherapy;
2. Patients with other malignancies, except basal cell carcinoma and carcinoma in situ..
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
6. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Surufatinib.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) ≤ 40%.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
10. History of hypersensitivity to any active or inactive ingredient of Surufatinib or to drugs with a similar chemical structure or class to Surufatinib.
11. Patients who are allergic to paclitaxel or other drugs prepared with polyoxyethyl castor oil, carboplatin or other platinum containing compounds.Patients with contraindications of Chemotherapy .
12. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerable Dose (MTD) | up to 12 months
  Usually refers to the highest dose at which a subject's probability of developing DLT does not exceed the probability of target toxicity during the regime-specified DLT observation period.
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib Combine With Immunotherapy and Chemotherapy as second-line therapy to Advanced CRC, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  OS was calculated from the date of pharmacy to death from any cause.
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Liangjun Zhu, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (5):
- China (5):
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu